CLINICAL TRIAL: NCT04020510
Title: Standard Injections Versus Reduced Injections for Intravesical onabotulinumtoxinA for Treatment of Idiopathic and Neurogenic Overactive Bladder: a Randomized Trial
Brief Title: Standard Injections Versus Reduced Injections for Intravesical onabotulinumtoxinA Treatment of Overactive Bladder
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Angela DiCarlo-Meacham, Principal Investigator, Walter Reed National Military Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0232
Record Dates: First submitted 2019-07-11; First posted 2019-07-16 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — onabotulinum toxin A; Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard Injections (Active Comparator): For idiopathic overactive bladder, 100 units of onabotulinumtoxinA mixed in 10mL of injectable saline injected in 20 sites with 0.5mL per injection along the posterior wall of the bladder above the trigone. For neurogenic overactive bladder, 200 units of onabotulinumtoxinA mixed in 30mL of injectable saline injected in 30 sites with 1mL per injection along the posterior wall of the bladder above the trigone.
  Interventions: Drug: onaBoNT-A
- Reduced Injections (Experimental): For idiopathic overactive bladder, 100 units of onabotulinumtoxinA mixed in 10mL of injectable saline injected in 5 sites with 2mL per injection in an "X" configuration on posterior wall of the bladder above the trigone. For neurogenic overactive bladder, 200 units of onabotulinumtoxinA mixed in 10mL of injectable saline injected in 5 sites with 2mL per injection in an "X" configuration on posterior wall of the bladder above the trigone.
  Interventions: Drug: onaBoNT-A

INTERVENTIONS:
Drug: onaBoNT-A — Intradetrusor onabotulinumtoxinA in either the standard number of injections or a reduced number of injections
  Other Names: Botox

SUMMARY:
OnabotulinumtoxinA is an effective treatment for both idiopathic and neurogenic overactive bladder and was FDA approved for this indication in 2013. The standard technique for injecting onabotulinumtoxinA into the detrusor is mixing 100 units of onabotulinumtoxinA into 10mL of injectable normal saline and injecting 20 sites with 0.5mL in the posterior wall of hte bladder for idiopathic overactive bladder and mixing 200 units into 30mL and injecting 30 sites with 1mL for neurogenic overactive bladder. The purpose of this study is to compare the efficacy of a technique using a reduced number of injections with the same dosage of onabotulinumtoxinA to the standard technique. The hypothesis is that the reduced technique will not be inferior in terms of efficacy as the standard technique and that there will be a lower incidence of urinary tract infections and urinary retention requiring catheterization post-procedure.

DETAILED DESCRIPTION:
Overactive bladder has a large economic burden within the United States and internationally. Patients are often non-compliant with first and second line treatments for overactive bladder or find that they do not significantly improve symptoms. Intradetrusor onabotulinumtoxinA injection has been showed in many studies to significantly improve overactive bladder symptoms and quality of life in patients and was approved by the FDA for the treatment of overactive bladder in 2013.

Intradetrusor onabotulinumtoxinA injections are often performed in the office setting under local anesthesia. The standard technique for injecting onabotulinumtoxinA into the detrusor is mixing 100 units of onabotulinumtoxinA into 10mL of injectable normal saline and injecting 20 sites with 0.5mL in the posterior wall of hte bladder for idiopathic overactive bladder and mixing 200 units into 30mL and injecting 30 sites with 1mL for neurogenic overactive bladder. Despite instillation of local anesthetic into the bladder prior to the procedure, many patients still find the procedure uncomfortable and may elect not to have treatment or to undergo treatment under sedation.

Some literature exists that suggests that a fewer number of injections with the same dosage of onabotulinumtoxinA still provides significant improvement in symptoms for patients with the potential for fewer adverse events, specifically urinary tract infection and urinary retention requiring catheterization.

The purpose of this study is to directly compare the standard techniqe for intradetrusor onabotulinumtoxinA injections to a reduced injection technique to compare efficacy and rates of adverse events between the two groups. The hypothesis is that the reduced injection technique will be non-inferior to the standard technique.

Participants in the study will be randomized to either the standard technique or the reduced technique at the time of their procedures, provided they meet the inclusion and exclusion criteria and provide written consent to participate. Efficacy will be measured using a series of validated patient questionnaires. Scores will be obtained at a baseline and then at two other time points post-procedure (4-12 weeks and 6-9 months). Rates of adverse outcomes, specifically urinary tract infection and urinary retention requiring catheterization, will also be obtained following the procedure.

Other than the randomization of patients into study and control groups and having patients complete a series of questionnaires, the care of patients undergoing intradetrusor onabotulinumtoxinA injections will follow the standard of care. All patients will be screened for urinary tract infection prior to the procedure and if they screen positive will have their procedures delayed until after they are treated. All patients will receive pre-procedure antibiotics according to the American Urological Association guidelines. All patients will be screened for urinary retention and for symptoms of urinary tract infection at their initial post-procedure follow-up at 4-12 weeks and treated accordingly if they develop either.

ELIGIBILITY:
Inclusion Criteria:

* Males or Females ≥ 18 years of age
* Predominant complaint of urinary urgency, urinary frequency or urge incontinence
* Failed at least one medication (inadequate or poorly tolerated response) or behavior modification technique (timed voiding, pelvic floor physical therapy, etc.), or decline such interventions
* Willingness to perform self-catheterization in the event of symptomatic urinary retention
* Ability to follow study instructions and likely to complete all required follow-up

Exclusion Criteria:

* Concurrent use of oral medications for treatment of OAB (anticholinergics or beta 3 agonists).
* Post void residual volume > 200 ml
* Symptomatic prolapse > POP-Q (Pelvic Organ Prolapse Quantification) stage 2 or greater that is untreated
* Evidence of active UTI (bladder infection)
* Any previous use of intradetrusor botulinum toxin (onabotulinumtoxinA or abobotulinumtoxinA) within the preceding 6 months
* Use of >/= 400 units bontulinum toxin in the preceding 3months in other areas of the body
* Procedure performed in the main operating room (not outpatient setting)
* Concurrent diagnosis of interstitial cystitis/painful bladder syndrome
* Females who are pregnant or planning a pregnancy during the study or who think that they may be pregnant at the start of the study, or females of childbearing potential who are unable or unwilling to use a reliable form of contraception during the study.
* Any medical condition that may put the subject at increased risk with exposure to botulinum-A toxin, including diagnosed myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis/motor neuron disease, neuropathy, renal stones, or any other disorder that might interfere with neuromuscular function
* Known allergy or sensitivity to any of the components of onabotulinumtoxinA
* Concurrent participation in another investigational drug or device study that could impact the results
* Any condition or situation that, in the investigator's opinion, may put the subject at significant risk, confound the study results, or interfere significantly with the subject's participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in overactive bladder symptom severity and health related quality of life scores on the overactive bladder questionnaire short form | 4-12 weeks post-procedure
  The overactive bladder questionnaire short form is a validated questionnaire assessing both symptoms and quality of life related to overactive bladder. The survey has two subscales, a health related quality of life scale and a symptom severity scale. Each subscale is scored separately with a range of 0 to 100. For health related quality of life a score of 0 indicates worst quality of life and 100 indicating best quality of life. For symptom severity, the scores also range from 0 to 100 but with higher scores indicating greater symptom severity and lower scores less symptom severity.
Mean change from baseline in overactive bladder symptom severity and health related quality of life scores on the overactive bladder questionnaire short form | 6-9 months post-procedure
  The overactive bladder questionnaire short form is a validated questionnaire assessing both symptoms and quality of life related to overactive bladder. The survey has two subscales, a health related quality of life scale and a symptom severity scale. Each subscale is scored separately with a range of 0 to 100. For health related quality of life a score of 0 indicates worst quality of life and 100 indicating best quality of life. For symptom severity, the scores also range from 0 to 100 but with higher scores indicating greater symptom severity and lower scores less symptom severity.
Mean change from baseline in overactive bladder symptoms on the International Consultation on Incontinence Questionnaire short form | 4-12 weeks post-procedure
  The International Consultation on Incontinence Questionnaire short form is a validated questionnaire assessing symptoms of overactive bladder and effect on quality of life. The scores range from 0 to 21 with higher scores indicating worse symptom severity and effect on quality of life.
Mean change from baseline in overactive bladder symptoms on the International Consultation on Incontinence Questionnaire short form | 6-9 months post-procedure
  The International Consultation on Incontinence Questionnaire short form is a validated questionnaire assessing symptoms of overactive bladder and effect on quality of life. Scores range from 0 to 21 with higher scores indicating greater symptom severity.
Mean change from baseline in overactive bladder symptoms assessed with the Patient Global Impression of Severity and Improvement scores | baseline, 4-12 weeks post-procedure and 6-9 months post-procedure
  The Patient Global Impression of Severity and Patient Global Impression of Improvement scores are validated single question surveys that assess patients' impression of the severity of their illness prior to treatment intervention and the degree of improvement following treatment intervention. The Patient Global Impression of Severity is a 4 point Likert scale ranging from 1 to 4 with 1 being normal and 4 being severe symptoms (mild and moderate completing the range of scores). The Patient Global Impression of Improvement is a 7 point Likert scale with 1 being very much better and 7 being very much worse (much better, a little better, no change, a little worse, and much worse completing the range of scores).
Mean change from baseline in overactive bladder symptoms assessed with the Patient Global Impression of Severity and Improvement scores | 4-12 weeks post-procedure
  The Patient Global Impression of Severity and Patient Global Impression of Improvement scores are validated single question surveys that assess patients' impression of the severity of their illness prior to treatment intervention and the degree of improvement following treatment intervention. The Patient Global Impression of Severity is a 4 point Likert scale ranging from 1 to 4 with 1 being normal and 4 being severe symptoms (mild and moderate completing the range of scores). The Patient Global Impression of Improvement is a 7 point Likert scale with 1 being very much better and 7 being very much worse (much better, a little better, no change, a little worse, and much worse completing the range of scores).
Mean change from baseline in overactive bladder symptoms and incontinence episodes using patient reported pad counts and episodes of nocturia | 6-9 months post-procedure
  Number of pads used for urge incontinence and nocturia episodes are frequent metrics used for assessing efficacy of overactive bladder treatments

SECONDARY OUTCOMES:
Incidence of urinary tract infection | 1 day to 12 weeks post-procedure
  Urinary tract infection is a common complication from intradetrusor onabotulinumtoxinA treatment
Incidence of urinary retention requiring intermittent catheterization | 2-6 weeks post-procedure
  Urinary retention is a common complication following intradetrusor onabotulinumtoxinA treatment
Mean change in pain from baseline following intradetrusor onabotulinumtoxinA injection using visual analog scale | immediately post-procedure
  Visual Analog Scales are validated tools for assessing pain. The scale is scored from 0 to 10 with 0 being no pain and 10 being worst possible pain.

CONTACTS AND LOCATIONS:
Overall Officials: Angela DiCarlo-Meacham, MD, Principal Investigator — Walter Reed National Military Medical Center
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Avallone MA, Sack BS, El-Arabi A, Guralnick ML, O'Connor RC. Less is more-A pilot study evaluating one to three intradetrusor sites for injection of OnabotulinumtoxinA for neurogenic and idiopathic detrusor overactivity. Neurourol Urodyn. 2017 Apr;36(4):1104-1107. doi: 10.1002/nau.23052. Epub 2016 Jun 10. PMID 27283922
- [Background] Lopez Ramos H, Torres Castellanos L, Ponce Esparza I, Jaramillo A, Rodriguez A, Moreno Bencardino C. Management of Overactive Bladder With OnabotulinumtoxinA: Systematic Review and Meta-analysis. Urology. 2017 Feb;100:53-58. doi: 10.1016/j.urology.2016.10.026. Epub 2016 Oct 24. PMID 27789302
- [Background] Sirls LT, Tennstedt S, Brubaker L, Kim HY, Nygaard I, Rahn DD, Shepherd J, Richter HE. The minimum important difference for the International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form in women with stress urinary incontinence. Neurourol Urodyn. 2015 Feb;34(2):183-7. doi: 10.1002/nau.22533. Epub 2013 Nov 23. PMID 24273137
- [Background] Yalcin I, Bump RC. Validation of two global impression questionnaires for incontinence. Am J Obstet Gynecol. 2003 Jul;189(1):98-101. doi: 10.1067/mob.2003.379. PMID 12861145
- [Background] Visco AG, Brubaker L, Richter HE, Nygaard I, Paraiso MF, Menefee SA, Schaffer J, Lowder J, Khandwala S, Sirls L, Spino C, Nolen TL, Wallace D, Meikle SF; Pelvic Floor Disorders Network. Anticholinergic therapy vs. onabotulinumtoxina for urgency urinary incontinence. N Engl J Med. 2012 Nov 8;367(19):1803-13. doi: 10.1056/NEJMoa1208872. Epub 2012 Oct 4. PMID 23036134
- [Background] Coyne KS, Matza LS, Thompson CL, Kopp ZS, Khullar V. Determining the importance of change in the overactive bladder questionnaire. J Urol. 2006 Aug;176(2):627-32; discussion 632. doi: 10.1016/j.juro.2006.03.088. PMID 16813906
- [Background] Ramirez-Castaneda J, Jankovic J, Comella C, Dashtipour K, Fernandez HH, Mari Z. Diffusion, spread, and migration of botulinum toxin. Mov Disord. 2013 Nov;28(13):1775-83. doi: 10.1002/mds.25582. Epub 2013 Jul 18. PMID 23868503
- [Background] Coelho A, Cruz F, Cruz CD, Avelino A. Spread of onabotulinumtoxinA after bladder injection. Experimental study using the distribution of cleaved SNAP-25 as the marker of the toxin action. Eur Urol. 2012 Jun;61(6):1178-84. doi: 10.1016/j.eururo.2012.01.046. Epub 2012 Feb 1. PMID 22306320
- [Background] Karsenty G, Denys P, Amarenco G, De Seze M, Game X, Haab F, Kerdraon J, Perrouin-Verbe B, Ruffion A, Saussine C, Soler JM, Schurch B, Chartier-Kastler E. Botulinum toxin A (Botox) intradetrusor injections in adults with neurogenic detrusor overactivity/neurogenic overactive bladder: a systematic literature review. Eur Urol. 2008 Feb;53(2):275-87. doi: 10.1016/j.eururo.2007.10.013. Epub 2007 Oct 16. PMID 17988791
- [Background] Liao CH, Chen SF, Kuo HC. Different number of intravesical onabotulinumtoxinA injections for patients with refractory detrusor overactivity do not affect treatment outcome: A prospective randomized comparative study. Neurourol Urodyn. 2016 Aug;35(6):717-23. doi: 10.1002/nau.22780. Epub 2015 Apr 24. PMID 25914349
- [Background] Stewart WF, Van Rooyen JB, Cundiff GW, Abrams P, Herzog AR, Corey R, Hunt TL, Wein AJ. Prevalence and burden of overactive bladder in the United States. World J Urol. 2003 May;20(6):327-36. doi: 10.1007/s00345-002-0301-4. Epub 2002 Nov 15. PMID 12811491
- [Background] Tijnagel MJ, Scheepe JR, Blok BF. Real life persistence rate with antimuscarinic treatment in patients with idiopathic or neurogenic overactive bladder: a prospective cohort study with solifenacin. BMC Urol. 2017 Apr 13;17(1):30. doi: 10.1186/s12894-017-0216-4. PMID 28403849
- [Background] Coyne KS, Thompson CL, Lai JS, Sexton CC. An overactive bladder symptom and health-related quality of life short-form: validation of the OAB-q SF. Neurourol Urodyn. 2015 Mar;34(3):255-63. doi: 10.1002/nau.22559. Epub 2014 Jan 13. PMID 25783168
- [Background] Crowner BE, Torres-Russotto D, Carter AR, Racette BA. Systemic weakness after therapeutic injections of botulinum toxin a: a case series and review of the literature. Clin Neuropharmacol. 2010 Sep-Oct;33(5):243-7. doi: 10.1097/WNF.0b013e3181f5329e. PMID 20852412

DOCUMENTS (1):
  • Informed Consent Form (2019-06-28): https://cdn.clinicaltrials.gov/large-docs/10/NCT04020510/ICF_000.pdf